CLINICAL TRIAL: NCT01892943
Title: Leber Hereditary Optic Neuropathy (LHON) Historical Case Record Survey
Status: Completed | Type: Observational
Sponsor: Santhera Pharmaceuticals (Industry)
Collaborators: European Vision Institute Clinical Research Network (Network)
Responsible Party: Sponsor
Other Study IDs: LHON HCR
Record Dates: First submitted 2013-06-26; First posted 2013-07-08 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2014-05

CONDITIONS: Leber Hereditary Optic Neuropathy (LHON)
MeSH Terms: conditions — Optic Atrophy, Hereditary, Leber

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Patients with LHON

SUMMARY:
The objective of this survey is to establish the clinical course of vision loss and recovery in patients with a genetically confirmed diagnosis of Leber Hereditary Optic Neuropathy (LHON).

Visual acuity changes over time from onset of symptoms and from visual acuity nadir will be the main endpoint analysed.

The survey will collect historically documented visual acuity data for all patients at participating sites with a genetically confirmed diagnosis of LHON. No exclusion criteria apply. Patients are not required to attend the clinic for the survey.

Data will be collected in a completely anonymous manner. Ethical approvals and data release agreements will be obtained as required by local regulations.

ELIGIBILITY:
Inclusion Criteria:

* patients with genetically confirmed diagnosis of LHON

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with genetically confirmed diagnosis of LHON
Sampling Method: Non-Probability Sample
Enrollment: 306 (Actual)
Dates: Start 2013-08; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Visual acuity | average 0 to 10 years (retrospective)
  The Entire duration of the disease patient by patient basis up to the date of completion of the Case Report Form (CRF).

CONTACTS AND LOCATIONS:
Overall Officials: Jose-Alain Sahel, MD, Principal Investigator — Centre de Recherche Institut de la Vision INSERMN
Locations (8):
- University Hospitals Leuven, Leuven, Belgium
- Glostrup Hospital/National Eye Clinic of the Kennedy Center/University of Copenhagen Department of Ophthalmology, Glostrup Municipality, Denmark
- France (2):
  - CHU Bordeaux, Bordeaux
  - CIC/CMR CHNO des Quinze-Vingts, Paris
- Italy (3):
  - Universty of Bari, Bari
  - Fondazione G.B. Bietti, Rome
  - San Raffaele Hospital, Segrate
- University Eye Clinic, Ljubljana, Slovenia